CLINICAL TRIAL: NCT00156481
Title: Smoking Practices Among Parents of Urban Children With Asthma: A Qualitative Study
Brief Title: A Qualitative Study About Smoking Practices
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Halcyon Hill Foundation (Other); Rochester City School District (Unknown); The Children's Institute (Other)
Responsible Party: Jill S. Halterman, MD, MPH, Halcyon Hill Foundation
Other Study IDs: 10095
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
This study involves in-depth interviews with parents of urban children with asthma and focus groups with additional parents in order to understand their attitudes and beliefs about smoking.

ELIGIBILITY:
Inclusion Criteria:

* Child with asthma
* Parents being current smokers, ex-smokers, or non-smokers

Exclusion Criteria:

* Non-English speaking families

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Parents of children with asthma in Rochester, NY
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2004-12; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Halterman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- Rochester - Families Homes, Rochester, New York, United States

REFERENCES:
- [Result] Halterman JS, Fagnano M, Conn KM, Lynch KA, DelBalso MA, Chin NP. Barriers to reducing ETS in the homes of inner-city children with asthma. J Asthma. 2007 Mar;44(2):83-8. doi: 10.1080/02770900601180545. PMID 17454320